CLINICAL TRIAL: NCT01359527
Title: A Dual Energy X-Ray Absorptiometry Comparison Of Periprosthetic Bone Loss Between Patients Undergoing Hip Resurfacing Surgery And Total Hip Arthroplasty
Brief Title: Dual Energy X-ray Absorptiometry (DXA) Comparison Hip Resurfacing Versus Total Hip Arthroplasty (THA)
Status: Completed | Type: Observational
Sponsor: Spokane Joint Replacement Center (Other)
Responsible Party: Principal Investigator, David F. Scott, MD, PI, Spokane Joint Replacement Center
Other Study IDs: SJRC-RSRF
Record Dates: First submitted 2011-05-22; First posted 2011-05-24 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis, Hip
Keywords: Total Hip Replacement; Hip Resurfacing; Femoral Remodeling; Bone Loss; Bone Mineral Density; BMD; DXA; DEXA; THA
MeSH Terms: conditions — Osteoarthritis, Hip; Bone Diseases, Metabolic | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hip Resurfacing
  Interventions: Device: Hip Resurfacing
- Total Hip Arthroplasty
  Interventions: Device: Total Hip Arthroplasty

INTERVENTIONS:
Device: Hip Resurfacing
  Groups: Hip Resurfacing
Device: Total Hip Arthroplasty
  Groups: Total Hip Arthroplasty

SUMMARY:
This study compares the change (loss) of bone mineral density (BMD) that occurs in the proximal femur after hip resurfacing and total hip replacement.

DETAILED DESCRIPTION:
This study compares the change (loss) of bone mineral density (BMD) that occurs in the proximal femur after hip resurfacing and total hip replacement. The goal is to evaluate the bone loss in the proximal femur resulting from hip resurfacing surgery and to compare this to the bone loss in the proximal femur resulting from total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 20 years
* Osteoarthritis
* Elective Total Hip Arthroplasty / Resurfacing
* Signed Informed Consent

Exclusion Criteria:

* Osteoporosis
* Revisions
* Femoral dysplasia
* Trochanteric osteotomy
* Inflammatory arthritis
* Breast-feeding, pregnancy, or women of child-bearing potential without documentation of a negative pregnancy test and not utilizing contraception
* Patients with a history of having taken or currently taking PTH, fluoride therapy or strontium ranelate or patients taking other chronic medications that in the Investigator's opinion are known to affect bone mineral density in a substantial way
* Patients with severe medical condition(s) that in the view of the Investigator prohibits participation in the study
* Use of any other investigational agent in the last 30 days

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing hip replacement or resurfacing for osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2008-12; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | Baseline, 6 weeks, 6 months, 1, 2, 3, 4, and 5 years post-operative
  To evaluate the bone loss in the proximal femur resulting from hip resurfacing surgery and to compare this to the bone loss in the proximal femur resulting from total hip arthroplasty.

SECONDARY OUTCOMES:
Harris Hip Score | Pre-operative, 6 weeks, 6 months, 1, 2, 3, 4, and 5 years post-operative
  Hip functional outcomes will be assessed using the Harris Hip Score

CONTACTS AND LOCATIONS:
Overall Officials: David Scott, MD, Principal Investigator — Spokane Joint Replacement Center
Locations (1):
- Spokane Joint Replacement Center, Spokane, Washington, United States